CLINICAL TRIAL: NCT01222715
Title: A Randomized Phase II Trial of Bevacizumab (Avastin) and Temsirolimus (Torisel) in Combination With Intravenous Vinorelbine and Cyclophosphamide in Patients With Recurrent/Refractory Rhabdomyosarcoma
Brief Title: Vinorelbine Tartrate and Cyclophosphamide in Combination With Bevacizumab or Temsirolimus in Treating Patients With Recurrent or Refractory Rhabdomyosarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02607; NCI-2011-02607 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); COG-ARST0921; CDR0000687113; ARST0921; ARST0921 (Other: Childrens Oncology Group); ARST0921 (Other: CTEP); U10CA098543 (NIH)
Record Dates: First submitted 2010-10-15; First posted 2010-10-18 (Estimated); Results first posted 2017-05-05 (Actual); Last update posted 2017-05-05 (Actual); Status verified 2017-03

CONDITIONS: Adult Rhabdomyosarcoma; Childhood Alveolar Rhabdomyosarcoma; Childhood Pleomorphic Rhabdomyosarcoma; Childhood Rhabdomyosarcoma With Mixed Embryonal and Alveolar Features; Previously Treated Childhood Rhabdomyosarcoma; Recurrent Adult Soft Tissue Sarcoma; Recurrent Childhood Rhabdomyosarcoma
MeSH Terms: conditions — Rhabdomyosarcoma; Sarcoma | interventions — Bevacizumab; Immunoglobulin G; Disulfides; Cyclophosphamide; temsirolimus; Sirolimus; Vinorelbine

ARMS (2):
- Arm I (vinorelbine tartrate, cyclophosphamide, bevacizumab) (Experimental): Patients receive vinorelbine tartrate IV over 6-10 minutes on days 1 and 8 and cyclophosphamide IV over 30-60 minutes on day 1. Patients also receive bevacizumab IV over 30-90 minutes on day 1.
  Interventions: Biological: Bevacizumab; Drug: Cyclophosphamide; Other: Laboratory Biomarker Analysis; Drug: Vinorelbine Tartrate
- Arm II (vinorelbine tartrate, cyclophosphamide, temsirolimus) (Experimental): Patients receive vinorelbine tartrate and cyclophosphamide as in arm I. Patients also receive temsirolimus IV over 30-60 minutes on days 1, 8, and 15.
  Interventions: Drug: Cyclophosphamide; Other: Laboratory Biomarker Analysis; Drug: Temsirolimus; Drug: Vinorelbine Tartrate

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF rhuMAb; Avastin; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF
  Arms: Arm I (vinorelbine tartrate, cyclophosphamide, bevacizumab)
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Temsirolimus — Given IV
  Other Names: CCI-779; CCI-779 Rapamycin Analog; Cell Cycle Inhibitor 779; Rapamycin Analog; Rapamycin Analog CCI-779; Torisel
  Arms: Arm II (vinorelbine tartrate, cyclophosphamide, temsirolimus)
Drug: Vinorelbine Tartrate — Given IV
  Other Names: Biovelbin; Eunades; KW-2307; Navelbine; Navelbine Ditartrate; NVB; Vinorelbine Ditartrate

SUMMARY:
This randomized phase II trial studies how well vinorelbine tartrate and cyclophosphamide work in combination with bevacizumab or temsirolimus in treating patients with recurrent or refractory rhabdomyosarcoma. Drugs used in chemotherapy, such as vinorelbine tartrate and cyclophosphamide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of rhabdomyosarcoma by blocking blood flow to the tumor. Temsirolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known whether combination chemotherapy is more effective when given together with bevacizumab or temsirolimus in treating rhabdomyosarcoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

l. To determine the feasibility of administering bevacizumab in combination with intravenous vinorelbine (vinorelbine tartrate) and cyclophosphamide (VC) in patients with recurrent rhabdomyosarcoma (RMS).

II. To determine the feasibility of administering temsirolimus in combination with VC in patients with recurrent RMS.

III. To estimate the event-free survival (EFS) of patients with recurrent/refractory RMS treated with bevacizumab and VC and compare with the EFS of those treated with temsirolimus and VC.

SECONDARY OBJECTIVES:

I. To estimate the initial (2 cycle) response rate of patients with recurrent/refractory RMS treated with bevacizumab and VC and compare with the response rate of those treated with temsirolimus and VC, and to also compare the best response rate on each regimen of protocol therapy.

II. To evaluate surrogate biological markers in patients with recurrent RMS and to estimate differences in these markers following treatment with bevacizumab and temsirolimus.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive vinorelbine tartrate intravenously (IV) over 6-10 minutes on days 1 and 8 and cyclophosphamide IV over 30-60 minutes on day 1. Patients also receive bevacizumab IV over 30-90 minutes on day 1.

ARM II: Patients receive vinorelbine tartrate and cyclophosphamide as in arm I. Patients also receive temsirolimus IV over 30-60 minutes on days 1, 8, and 15.

In both arms, treatment repeats every 21 days for 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up annually for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis

  * Patients with first relapse or progression of rhabdomyosarcoma are eligible
  * Patients with primary refractory disease are eligible

    * Primary refractory disease is defined as first progression after receiving at least one course of cyclophosphamide or ifosfamide containing chemotherapy without prior demonstration of a radiographic response to chemotherapy (progression on irinotecan-containing chemotherapy without cyclophosphamide or ifosfamide containing chemotherapy will not be considered a first progression)
  * Note: Patients without measurable or evaluable disease are eligible
* Patients must have had a previous histological verification of rhabdomyosarcoma at original diagnosis
* Patients must have a Karnofsky or Lansky performance status score of >= 50%, corresponding to Eastern Cooperative Oncology Group (ECOG) categories of 0, 1, or 2; use Karnofsky for patients > 16 years of age and Lansky for patients =< 16 years of age
* Patients must have a life expectancy of >= 8 weeks
* Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study
* Myelosuppressive chemotherapy: Must not have received within 3 weeks prior to entry onto this study (4 weeks if prior nitrosourea)
* Biologic (anti-neoplastic agent):

  * Patients may have received prior therapy with oral tyrosine kinase inhibitors or other similar agents; at least 7 days must have elapsed since the completion of therapy with a biologic agent and all toxicities must have resolved to < grade 2 prior to enrollment
  * 3 half-lives (or 6 weeks) must have elapsed since previous monoclonal antibody therapy prior to enrollment on this study
* Myeloid growth factor: Must not have received within 1 week prior to entry onto this study
* Radiation therapy (RT): At least 4 weeks must have elapsed between RT and study entry; previously radiated lesions cannot be used to assess response unless those sites are the sites of disease progression
* Stem cell transplant (SCT): For autologous SCT, >= 3 months must have elapsed; for allogeneic SCT, >= 6 months must have elapsed and no evidence of active graft vs. host disease
* Patients must have recovered from any surgical procedure before enrolling on this study

  * Minor surgical procedures (e.g., biopsies involving core or fine-needle aspiration procedures, infusaport or Broviac line placement, paracentesis, or thoracocentesis) need to have fully healed and occurred > 7 days prior to enrollment
  * Patients who have had a major surgical procedure (such as laparotomy, thoracotomy, open biopsy, or resection of tumor) can only be enrolled on study > 28 days from such procedure
* Peripheral absolute neutrophil count (ANC) >= 750/μL
* Platelet count >= 75,000/μL (transfusion independent, defined as without transfusion for >= 1 week prior to enrollment)
* Hemoglobin >= 8.0 g/dL (may receive packed red blood cells [PRBC] transfusions)
* Bone marrow disease involvement of tumor is allowed, however, peripheral blood count criteria must still be met
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 mL/min/1.73 m^2 OR a serum creatinine based on age/gender as follows:

  * =< 0.4 mg/dL (for patients aged 1 month to < 6 months)
  * =< 0.5 mg/dL (for patients aged 6 months to < 1 year)
  * =< 0.6 mg/dL (for patients aged 1 to < 2 years)
  * =< 0.8 mg/dL (for patients aged 2 to < 6 years)
  * =< 1 mg/dL (for patients aged 6 to < 10 years)
  * =< 1.2 mg/dL (for patients aged 10 to < 13 years)
  * =< 1.4 mg/dL (for female patients aged >= 13 years)
  * =< 1.5 mg/dL (for male patients aged 13 to < 16 years)
  * =< 1.7 mg/dL (for male patients aged >= 16 years)
* Urine protein level:

  * Patients aged =< 17 years: Urine protein to creatinine (UPC) ratio should be calculated; UPC ratio must be =< 1 for patient to be eligible
  * Patients aged > 17 years: Urine protein should be screened by urine analysis; if protein is 2+ or higher, 24-hour urine protein must be obtained and the level must be < 1,000 mg for patient enrollment
* Total bilirubin =< 1.5 x upper limit of normal (ULN) for age
* Shortening fraction of >= 27% by echocardiogram or ejection fraction of >= 50% by radionuclide angiogram

Exclusion Criteria:

* Patients with botryoid histology, any stage or group, are ineligible
* Patients with embryonal histology, stage I or clinical group 1 at initial disease presentation, who present with local or regional recurrence, are ineligible
* Patients who previously received craniospinal irradiation are ineligible
* Patients who previously received vinorelbine, bevacizumab, temsirolimus, or any other direct vascular endothelial growth factor (VEGF)/vascular endothelial growth factor receptor (VEGFR-) or mammalian target of rapamycin (mTOR-) targeting agents are ineligible
* Patients with known central nervous system (CNS) disease (excluding intracranial/intraspinal extension secondary to local progression of a parameningeal or paraspinal primary), except for those with treated brain metastasis, are ineligible

  * Treated brain metastases are defined as having no ongoing requirement for steroids and no evidence of progression or hemorrhage after treatment for at least 3 months, as ascertained by clinical examination and brain imaging (magnetic resonance imaging [MRI] or computed tomography [CT]); stable dose of anticonvulsants are allowed; treatment for brain metastases may include whole-brain radiotherapy (WBRT), radiosurgery (RS; Gamma Knife, linear accelerator [LINAC], or equivalent), or a combination as deemed appropriate by the treating physician
  * Patients with CNS metastases treated within 3 months prior to enrollment by neurosurgical resection or brain biopsy are ineligible
* Patients who receive radiation or chemotherapy (inclusive of palliative intent) for first disease progression or relapse of rhabdomyosarcoma prior to enrollment are ineligible
* Female patients who are pregnant are ineligible
* Lactating females are not eligible unless they have agreed to discontinue breastfeeding
* Female patients of childbearing potential are not eligible unless a negative pregnancy test result has been obtained
* Sexually active patients of reproductive potential are not eligible unless they have agreed to use an effective contraceptive method for the duration of their study participation
* Patients with a documented chronic non-healing wound, ulcer, or significant trauma injury (those with bone fractures, including pathological fractures, or requiring surgical intervention) within 28 days prior to beginning therapy are ineligible
* Patients with evidence of intratumoral hemorrhage, gastrointestinal bleeding, or on anticoagulation for thrombosis or history of thrombosis are ineligible
* Patients with uncontrolled hypertension are ineligible; uncontrolled hypertension is defined as follows:

  * Patients aged =< 17 years: greater than 95th percentile systolic and diastolic blood pressure based on age and height that is not controlled by one antihypertensive medication
  * Patients aged > 17 years: systolic blood pressure >= 160 mm Hg and/or diastolic blood pressure >= 90 mm Hg that is not controlled by one antihypertensive medication
* Patients currently taking anticoagulants or antiplatelet agents with the exception of aspirin (=< 81 mg/day) are ineligible
* Patients with history of central venous catheter (CVC)-associated thrombosis requiring systemic anticoagulation are ineligible; Note: Patients with history of sluggish flow from CVC or CVC-associated thrombosis treated with tissue plasminogen activator (TPA) only are not excluded
* Patients with clinically significant cardiovascular disease are excluded:

  * History of cerebrovascular accident (CVA) within the prior 6 months
  * Myocardial infarction or unstable angina within the prior 6 months
  * New York Heart Association grade 2 or greater congestive heart failure
  * Serious and inadequately controlled cardiac arrhythmia
  * Significant vascular disease (e.g., aortic aneurysm, history of aortic dissection)
  * Clinically significant peripheral vascular disease
* Patients diagnosed with rhabdomyosarcoma as a second malignant neoplasm are not eligible
* Patients with history of any second malignant neoplasm who have received chemotherapy or radiation for the treatment of that malignancy are not eligible

Max Age: 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 87 (Actual)
Dates: Start 2010-10; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leo Mascarenhas, Principal Investigator — Children's Oncology Group
Locations (184):
- United States (163):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Southern California Permanente Medical Group, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Children's Hospital Central California, Madera, California
  - Children's Hospital and Research Center at Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Lee Memorial Health System, Fort Myers, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Florida Hospital Orlando, Orlando, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - UF Cancer Center at Orlando Health, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Hospital, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Memorial University Medical Center, Savannah, Georgia
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Riley Hospital for Children, Indianapolis, Indiana
  - Saint Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Kosair Children's Hospital, Louisville, Kentucky
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Floating Hospital for Children at Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Michigan State University Clinical Center, East Lansing, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Kalamazoo Center for Medical Studies, Kalamazoo, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - The Childrens Mercy Hospital, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Winthrop University Hospital, Mineola, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Columbia University/Herbert Irving Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Mission Hospital-Memorial Campus, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Medical Center-Fargo, Fargo, North Dakota
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - The Toledo Hospital/Toledo Children's Hospital, Toledo, Ohio
  - Mercy Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at Saint Francis, Tulsa, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Hershey Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Palmetto Health Richland, Columbia, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Greenville Cancer Treatment Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Texas Tech University Health Science Center-Amarillo, Amarillo, Texas
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont College of Medicine, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Childrens Hospital-King's Daughters, Norfolk, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - West Virginia University Charleston, Charleston, West Virginia
  - Saint Vincent Hospital, Green Bay, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Australia (3):
  - Sydney Children's Hospital, Randwick, New South Wales
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Princess Margaret Hospital for Children, Perth, Western Australia
- Canada (16):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Child Health Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Chedoke Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston General Hospital, Kingston, Ontario
  - Children's Hospital, London, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - The Montreal Children's Hospital of the MUHC, Montreal, Quebec
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Québec, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- New Zealand (2):
  - Starship Children's Hospital, Grafton, Auckland
  - Christchurch Hospital, Christchurch

REFERENCES:
- [Derived] Mascarenhas L, Chi YY, Hingorani P, Anderson JR, Lyden ER, Rodeberg DA, Indelicato DJ, Kao SC, Dasgupta R, Spunt SL, Meyer WH, Hawkins DS. Randomized Phase II Trial of Bevacizumab or Temsirolimus in Combination With Chemotherapy for First Relapse Rhabdomyosarcoma: A Report From the Children's Oncology Group. J Clin Oncol. 2019 Nov 1;37(31):2866-2874. doi: 10.1200/JCO.19.00576. Epub 2019 Sep 12. PMID 31513481

RESULTS

PARTICIPANT FLOW:
Groups:
- Regimen A: The cyclophosphamide plus vinorelbine combination was administered at 1.2 g/m2 every 3 weeks and 25 mg/m2/dose (administered weekly on the first 2 out of every 3 weeks), respectively. Bevacizumab was administered at 15 mg/kg every 3 weeks.
- Regimen B: The cyclophosphamide plus vinorelbine combination was administered at 1.2 g/m2 every 3 weeks and 25 mg/m2/dose (administered weekly on the first 2 out of every 3 weeks), respectively. Temsirolimus was administered at 15 mg/m2/week intravenously.
Period: Overall Study
Arm/Group | Regimen A | Regimen B
Started | 44 | 43
Completed | 8 | 16
Not Completed | 36 | 27
Not completed — Adverse Event | 0 | 4
Not completed — Death | 0 | 1
Not completed — Lack of Efficacy | 22 | 14
Not completed — Physician Decision | 12 | 2
Not completed — Refusal of further protocol therapy | 0 | 4
Not completed — Pt cannot receive treatment for >9 wks | 1 | 1
Not completed — Ineligible | 0 | 1
Not completed — Surgery or radiation therapy in 1st 6 wk | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Regimen A | Regimen B | Total
Number analyzed (Participants) | 44 | 43 | 87
Age, Continuous [Mean (Standard Deviation); unit: Months] | 116.35 (72.82) | 140.65 (75.93) | 128.36 (74.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 20 | 42
  Male | 22 | 23 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 10 | 19
  Not Hispanic or Latino | 35 | 31 | 66
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 7 | 7 | 14
  White | 30 | 27 | 57
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 7 | 12

OUTCOME MEASURES:

1. Primary Outcome: Event Free Survival Probability
Description: Probability of no relapse, secondary malignancy, or death after 1 year in the study.
Time Frame: 1 year
Population: Only eligible participants were analyzed.
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Regimen A | Regimen B
Number analyzed (Participants) | 44 | 42
Probability | 0.23 [0.10 to 0.35] | 0.43 [0.28 to 0.58]
Statistical Analysis 1: Comparison: Regimen A vs Regimen B; The event free survival distributions of patients in Regimen A and Regimen B were compared using the log-rank test; Test type: Superiority or Other; p = 0.0124, Log Rank

2. Primary Outcome: Rate of Dose-Limiting Toxicities
Description: The following events will be considered dose-limiting toxicities (DLTs): Toxicity causing delays > 14 days in delivery of a 21-day cycle of therapy; Grade ≥ 3 mucositis > 3 days duration; Grade ≥ 3 thromboembolic events; Grade ≥ 3 bleeding events; Grade ≥ 3 pulmonary events; Grade ≥ 3 hypertension; Grade 3 hyperglycemia (uncontrolled); Grade ≥ 4 hyperglycemia; Grade ≥ 4 hyperlipidemia (including cholesterol and triglycerides) that does not return to ≤ Grade 2 levels with appropriate medical management within 35 days; Grade ≥ 2 perforation including fistula or leak (gastrointestinal or any other organ); Grade ≥ 3 proteinuria; Grade ≥ 3 cardiac toxicity; Grade ≥ 3 intra-abdominal abscess/infection; Grade ≥ 3 wound complication (wound infection or dehiscence); Grade ≥ 1 Reversible Posterior Leukoencephalopathy Syndrome (RPLS); Grade ≥ 1 Microangiopathy, or Hemolytic-uremic syndrome (HUS) or Thrombotic thrombocytopenic Purpura (TTP).
Time Frame: From the date of randomization until a maximum of 12 cycles (21 days per cycle) of treatment in the absence of disease progression or unacceptable toxicities.
Population: Only eligible participants were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Regimen A | Regimen B
Number analyzed (Participants) | 44 | 42
Percentage of participants | 2 [0 to 7] | 21 [9 to 34]

3. Secondary Outcome: Response Rate (CR + PR)
Description: Complete or partial anatomical response rate. Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. Overall Response (OR) = CR + PR.
Time Frame: From the date of randomization until a maximum of 2 cycles (21 days per cycle) of treatment in the absence of disease progression or unacceptable toxicities.
Population: Only eligible participants with overall response evaluated were analyzed.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Regimen A | Regimen B
Number analyzed (Participants) | 40 | 38
Proportion of participants | 0.3250 [0.1799 to 0.4701] | 0.4737 [0.3149 to 0.6324]

4. Other Pre Specified Outcome: Biomarker Levels
Description: Biomarker data will be summarized for each response category, at each time point using either means and standard deviations or medians and ranges.
Time Frame: Up to 36 weeks
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Changes in Angiogenesis-associated Plasma Markers Between Patients by Treatment
Description: First, the distributions of these markers will be compared at 'end of 2 cycles' between treatments using a 2-independent sample non-parametric test. The mean will also be modeled for each of these markers (or a transformation of the marker to near normality) as a function of time and treatment using GEEs which are designed to take into account the internal correlation of repeated measurements taken on the same subject. Associations between progression-free survival and changes in each of the biomarkers will be investigated using univariate Cox proportional hazards regression analysis.
Time Frame: Baseline up to day 42
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Clinical Predictors, Including Histologic and Molecular Subtype, Age, Stage, and Site
Description: These known risk factors will be compared to genomic features like gene and ribonucleic acid (RNA) expression values, as well as combinations of the two and splice variants of known genes, in order to identify those features most related to treatment resistance and poor outcome (overall survival and failure-free survival) using a Cox proportional hazards model of gene expression with cross validation.
Time Frame: Up to 5 years
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Clinical Response
Description: The data reported in 2 groups will be summarized using numbers and percentages of patients in each stratum and at each time point (baseline, after course 2, at the time of best response and end of therapy or progressive disease, whichever comes first). A binomial generalized estimating equation (GEE) model will be fitted to the data. The variables in the model will be time, treatment group and a biomarker. The beta coefficient of the biomarker will quantify the strength of the association between clinical response and the biomarker, beyond the association of the outcome to the other variables.
Time Frame: Up to 5 years
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Levels of Biomarkers Related to the Effect of Temsirolimus on the Unfolded Protein Response
Time Frame: Up to 36 weeks
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Progression-free Survival
Description: Progression-free survival data will be explored using Kaplan Meier analysis. Associations between this outcome and each of the biomarkers will be investigated using univariate Cox proportional hazards regression analysis.
Time Frame: Up to 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Groups:
- Regimen A: Vinorelbine/cyclophosphamide (VC) + bevacizumab
- Regimen B: Vinorelbine/cyclophosphamide (VC) + temsirolimus
Arm/Group | Regimen A | Regimen B
Serious Adverse Events (participants affected / at risk) | 35/44 | 32/42
Other Adverse Events (participants affected / at risk) | 28/44 | 30/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regimen A (N=44) | Regimen B (N=42)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Catheter related infection (Infections and infestations) | 0 (0) | 1 (1)
CPK increased (Investigations) | 0 (0) | 1 (1)
Death NOS (General disorders) | 27 (27) | 15 (15)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 3 (4)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (2)
Ejection fraction decreased (Investigations) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Esophageal infection (Infections and infestations) | 0 (0) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (7) | 9 (15)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 4 (6)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Leukemia secondary to oncology chemotherapy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 6 (6)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 7 (7)
Neutrophil count decreased (Investigations) | 0 (0) | 2 (2)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 3 (3) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (4) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 1 (1)
Typhlitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Weight loss (Investigations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regimen A (N=44) | Regimen B (N=42)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 4 (4)
Activated partial thromboplastin time prolonged (Investigations) | 2 (2) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 5 (8)
Alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 7 (8) | 8 (8)
Anorexia (Metabolism and nutrition disorders) | 2 (3) | 2 (2)
Anxiety (Psychiatric disorders) | 2 (2) | 3 (3)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 3 (4)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Cholesterol high (Investigations) | 1 (1) | 1 (1)
Conjunctivitis (Eye disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 1 (1)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Edema face (General disorders) | 0 (0) | 1 (1)
Ejection fraction decreased (Investigations) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Eyelid function disorder (Eye disorders) | 0 (0) | 1 (1)
Facial muscle weakness (Nervous system disorders) | 1 (1) | 0 (0)
Facial nerve disorder (Nervous system disorders) | 1 (1) | 0 (0)
Facial pain (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 7 (12) | 7 (20)
Fever (General disorders) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 5 (5) | 4 (6)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1) | 5 (5)
Hypoalbuminemia (Metabolism and nutrition disorders) | 7 (7) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (2) | 5 (10)
Hyponatremia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Ileus (Gastrointestinal disorders) | 1 (1) | 1 (2)
Infections and infestations - Other, specify (Infections and infestations) | 1 (2) | 0 (0)
INR increased (Investigations) | 1 (1) | 0 (0)
Investigations - Other, specify (Investigations) | 1 (1) | 0 (0)
Keratitis (Eye disorders) | 1 (1) | 0 (0)
Lymphedema (Vascular disorders) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 6 (11) | 6 (9)
Mucosal infection (Infections and infestations) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 2 (3)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 3 (12) | 4 (6)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Oculomotor nerve disorder (Nervous system disorders) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 6 (6) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pelvic infection (Infections and infestations) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 3 (3)
Photophobia (Eye disorders) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 6 (9) | 4 (8)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Renal calculi (Renal and urinary disorders) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Trismus (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 5 (10) | 5 (6)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less